CLINICAL TRIAL: NCT04440384
Title: Long Term Evaluation of Function and Quality of Life After Pollicisation
Acronym: Polliglobal
Status: Withdrawn | Type: Observational
Why Stopped: 0 INCLUSION
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0399
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Patients That Had Pollicization Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Functional evaluation — Patients will complete these forms and tests :
  Box and block test, Purdue peg board, Percival, Nine hole peg, T-GAP, EGF, MAHVIE, DASH, RAND36, CHQ-PF28, CHQ-CF45, CGI-S

SUMMARY:
The study aims at describing long term functional outcome of patients that underwent pollicisation surgery.

The hypothesis of the study is that there are prognostic factors of good function results of pollicisation (based on T-GAP classification for function) that will be searched on univariate and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* More than 7 years and less than 50 years
* Underwent unilateral or bilateral pollicisation surgery
* For children : non opposition of the parents
* For adults : non opposition

Exclusion Criteria:

- Patients able to understand the research and to answer to forms

Ages: 7 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient that underwent pollicisation surgery more than 5 years before
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
T-GAP score | At baseline, Day 0 (>5 years post-surgery)
  The Thumb Grasp and Pinch assessment (T-GAP) is a new outcome measure that classifies grasp and pinch styles to quantify use of the new thumb.
  Scoring is based on principles of hand development and skill using a 7-point hierarchical scale including abnormal (scores of 1e3) and normal (scores of 4e7) grasp patterns, with more mature patterns receiving higher points.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital femme mère enfant, Bron, France